CLINICAL TRIAL: NCT04800848
Title: Effects of the N95/FFP2 Face Mask on Physical Fitness in Children
Brief Title: Effects of the Face Mask on Physical Fitness in Children
Acronym: MaskFIT
Status: Completed | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Hugo Olmedillas Fernandez, Associate Professor, University of Oviedo
Other Study IDs: UO2021-01
Record Dates: First submitted 2021-03-09; First posted 2021-03-16 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Physical Fitness; Health; Childhood ALL; Emotional Stress; Sedentary Behavior; Cardiorespiratory Fitness
Keywords: Exercise; Alpha fitness battery; Kids; N95/FFP2; Physical Activity; CDI
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Stress, Psychological; Sedentary Behavior; Motor Activity | interventions — Masks

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mask/No Mask: The group will perform both situations in a randomized cross-over design:
  * 1. Scholars will perform the fitness test with the use of a N95/FFP2 face mask
  * 2. Scholars will perform the fitness test without the use of a N95/FFP2 face mask
  Interventions: Device: Mask

INTERVENTIONS:
Device: Mask — Physical Fitness is evaluated with the use of a face mask

SUMMARY:
The aim of this multicenter randomized crossover design study is to evaluate a sample of 500 boys and girls from public and private schools in the Principality of Asturias, aged between 6 and 12 years, with the objective of determining the level of physical condition, as well as to evaluate the effect of the use of FFP2/N95 face masks during the execution of the ALPHA Fitness battery, and the emotional effects caused by the use of these masks. This is a sample obtained by accessibility, in which the sampling will be stratified by age and academic year.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 and 12 years old.
2. Be able to perform all the tests and procedures that comprise the study.
3. Have signed informed parental consent.

Exclusion Criteria:

1. To take drugs that can affect the measurements
2. Contraindications or pathologies associated with exercise

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between 6 an 12 years that attend classes in state or private schools.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Physical Activity | at the beginning of the study (Day 1)
  The Physical Activity Questionnaire for Children (PAQ-C) will be administered to determine the amount and intensity of physical activity that children perform during a week. It consists of ten items, nine of which are used to calculate the activity level and the other item assesses whether any illness or other event prevented the child from doing regular activities in the last week. The overall result of the test is a score from 1 to 5, with higher scores indicating a higher level of activity.
Sedentarism | at the beginning of the study (Day 1)
  In order to know the sedentary behaviors of schoolchildren, a questionnaire will be passed to them that seeks to know the time they habitually dedicate to various sedentary behaviors. The questionnaire assess the amount of time spent doing 6 behaviors (watching television, playing computer, playing video games, surfing the Internet for hobby, surfing the Internet by study, sitting and studying). The 6 items were completed separately for weekdays and weekend days. With a scale from 1 to 7, such that higher scores indicate a higher level of sedentary lifestyle.
Emotional states | at the beginning of the study (Day 1)
  To evaluate the emotional state, the Children's Depression Inventory (CDI) questionnaire will be implemented, which consists of two scales: dysphoria (depressive mood, sadness, worry, etc.) and negative self-esteem (judgments of inefficiency, ugliness, badness, etc.) with which to measure the effects of the pandemic on the child population and the situation of anxiety that it produces. The questionnaire will be answered directly by the children, as a self-report.
  The original version has 27 items, with five subscales within the assessment that measure different components of depression, with three response options for each item.
Handgrip strength | at the beginning of the study (Day 1)
  The isometric strength of the upper body (manual grip) using a manual dynamometer with adjustable grip (Takei TKK-5401) and for this purpose there is a table-rule to adjust the grip according to the length of the subject's palm. The test will be performed twice, alternately with both hands, and the best result obtained will be recorded.
Horizontal Jump | at the beginning of the study (Day 1)
  The test will be carried out with or without face mask depending on the cross design.
  The horizontal jump with feet together measures the explosive strength of the lower body. Each student will perform the test twice and the best result obtained will be recorded. If in either of the two attempts the child falls backwards or contacts the surface with a part of the body other than the feet, a new jump will be allowed.
Horizontal Jump | Day 2 (two weeks later)
  Those who performed the first measurement with a face mask, in the second measurement will perform the test without a face mask, and vice versa.
  The horizontal jump with feet together measures the explosive strength of the lower body. Each student will perform the test twice and the best result obtained will be recorded. If in either of the two attempts the child falls backwards or contacts the surface with a part of the body other than the feet, a new jump will be allowed.
Speed and agility | at the beginning of the study (Day 1)
  The test will be carried out with or without face mask depending on the cross design.
  The 4 x 10m speed and agility test measures speed of movement, agility and coordination. Participants will perform the test twice, with the best result being recorded in seconds to one decimal place. The test will be performed on a non-slip surface so that there is no possibility of slipping.
Speed and agility | Day 2 (two weeks later)
  Those who performed the first measurement with a face mask, in the second measurement will perform the test without a face mask, and vice versa.
  The 4 x 10m speed and agility test measures speed of movement, agility and coordination. Participants will perform the test twice, with the best result being recorded in seconds to one decimal place. The test will be performed on a non-slip surface so that there is no possibility of slipping.
Aerobic capacity | at the beginning of the study (Day 1)
  The test will be carried out with or without face mask depending on the cross design.
  The 20m shuttle run test also known as 'Course Navette' is a maximal effort test that measures the maximum aerobic capacity, allowing to know the current and future cardiovascular health profile of the children who perform the study. The test will be performed once, over a uniform surface of 30 meters, 20 meters of which will be used for the test. When the child stops, the last stage or number announced by a CD with the test protocol will be recorded, which will set the pace to be followed throughout the test. The test will be executed individually as a preventive measure.
Aerobic capacity | Day 2 (two weeks later)
  Those who performed the first measurement with a face mask, in the second measurement will perform the test without a face mask, and vice versa.
  The 20m shuttle run test also known as 'Course Navette' is a maximal effort test that measures the maximum aerobic capacity, allowing to know the current and future cardiovascular health profile of the children who perform the study. The test will be performed once, over a uniform surface of 30 meters, 20 meters of which will be used for the test. When the child stops, the last stage or number announced by a CD with the test protocol will be recorded, which will set the pace to be followed throughout the test. The test will be executed individually as a preventive measure.
Comfort with the use of masks | at the beginning of the study (Day 1)
  The test will be carried out with or without face mask depending on the cross design. A visual scale which allow to measure the perception of the comfort level of the students with and without the N95/FFP2 face masks just after finished each test of the Alpha Fitness Battery. It is a visual scale from 0 to 10, ranging from comfortable, uncomfortable to extremely uncomfortable.
Comfort with the use of masks | Day 2 (two weeks later)
  Those who performed the first measurement with a face mask, in the second measurement will perform the test without a face mask, and vice versa.
  A visual scale which allow to measure the perception of the comfort level of the students with and without the N95/FFP2 face masks just after finished each test of the Alpha Fitness Battery. It is a visual scale from 0 to 10, ranging from comfortable, uncomfortable to extremely uncomfortable.
Height | at the beginning of the study (Day 1)
  Height is measured with a height rod to the nearest 0.1 cm (SECA 225, SECA, Hamburg, Germany),
Weight | at the beginning of the study (Day 1)
  Weight of the children is measured by a 0.1 kg precision bascule (SECA 861, SECA, Hamburg, Germany)
waist circumference | at the beginning of the study (Day 1)
  The waist circumference are measured following the ISAK protocol and measurement technique with an anthropometric tape (Holtain).

CONTACTS AND LOCATIONS:
Locations (1):
- Hugo Olmedillas, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No